CLINICAL TRIAL: NCT02414776
Title: Phase Ib/II Study of Hydroxychloroquine in Metastatic ER-Positive Breast Cancer Progressing on Hormonal Therapy
Brief Title: Hydroxychloroquine in Metastatic Estrogen Receptor-Positive Breast Cancer Progressing on Hormonal Therapy
Acronym: ABC01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI Leaving Site
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIRB 20140460
Record Dates: First submitted 2015-01-19; First posted 2015-04-13 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Estrogen Receptor Positive Breast Cancer
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hydroxychloroquine plus hormonal therapy (Experimental): Add hydroxychloroquine to the current hormonal therapy
  Interventions: Drug: hydroxychloroquine

INTERVENTIONS:
Drug: hydroxychloroquine — administration of hydroxychloroquine in combination with the current hormonal therapy
  Other Names: Plaquenil

SUMMARY:
To determine the safety and tolerability of orally administered hydroxychloroquine with hormonal therapy.

To assess the response rate of hydroxychloroquine in combination with hormonal therapy.

DETAILED DESCRIPTION:
To determine the number of patients with adverse effects

To assess the clinical response to the combination

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age with histologically confirmed, metastatic ER + breast cancer with clinical progression of disease (including radiographically stable disease with at least 50% increment of an elevated tumor marker by two measurements at least 2 weeks apart (this particular tumor marker will be used for disease status assessment in the study) on current hormonal therapy with PFS for at least 3 months.
2. Karnofsky Performance Status (KPS) ≥70% and a life expectancy >3 months.
3. Participants must have at least one target visceral lesion that allows for evaluation of tumor response or in the case of bone-only metastases, patients need to have a positive imaging study such as bone scan, magnetic resonance imaging (MRI) or positron emission tomography-computed tomography (PET-CT) or CT, and an elevated tumor marker at least twice as high as upper limit.
4. Absolute neutrophil count > 1500 mm3, platelet count ≥ 80×109 L, hemoglobin ≥ 8.5 g/dL
5. Creatinine clearance ≥ 30 mL/min, total bilirubin ≤ 2 mg/dL, AST/ALT ≤ 3 times the upper limit of normal range
6. No remaining grade 2 or higher toxicity from prior cancer therapies unless judged to be clinically insignificant by the Principal Investigator
7. At least two (2) weeks from prior major surgery
8. Willingness to provide permission to biopsy one of the lesions if applicable before the study (All the patients are encouraged to have post-therapy biopsy upon progression of disease, but it is optional) as well as blood samples for pertinent laboratory studies
9. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must be willing to use an acceptable non-hormonal contraceptive method (abstinence, or double barrier method) for the duration of the study and for 30 days following the last dose of study drug, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial -

Exclusion Criteria:

1. On combination hormonal therapy with everolimus or any other investigational agent
2. Patients have symptomatic untreated brain metastasis or leptomeningeal metastases or treated but still symptomatic requiring the use of steroid 18Jul2014 Protocol v3: ABC 01 Anti-Autophagy for Met Breast Cancer Page 4 of 16
3. Lymphangitic carcinomatosis involving ≥ 50% of the lungs; evidence of metastases involving more than one third of the liver on sonogram or computed tomography
4. Lactating females
5. Uncontrolled cardiac disease, congestive heart failure, angina or hypertension
6. Myocardial infarction or unstable angina within 2 months of treatment
7. Known human immunodeficiency virus (HIV) infection or chronic active Hepatitis B or C (patients are NOT required to be tested for the presence of such viruses prior to therapy on this protocol)
8. Active clinically serious infection > CTCAE (version 4.03) Grade 2
9. Serious non-healing wound, ulcer, or bone fracture
10. Concurrent psychiatric illness/social situations that would limit safety and compliance with study requirements
11. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements
12. Currently receiving any other investigational therapeutic agents
13. Patients with known glucose-6-phosphate dehydrogenase deficiency, porphyria, cirrhosis or any other conditions with potential significant known risks
14. Patients with history of retinal damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of the safety profile of orally administered hydroxychloroquine with hormonal therapy | 18 months
  Assess the dose-limiting side effects such as neutropenia, anemia, or thormbocytopenia, or non-hematologic side effects nausea, vomiting, diarrhea, or vision problems at the study dose

SECONDARY OUTCOMES:
The recommended phase 2 clinical dose (RP2D) of orally administered hydroxychloroquine with hormonal therapy | 18 months
  orally administered hydroxychloroquine with hormonal therapy
The pharmacodynamic (PD) profile of hydroxychloroquine with hormonal therapy | 18 months
  microtubule-associated protein 1 light chain 3 b (LC3b) level in the biopsy, WBCs in pre- and post-treatment samples
The anti-tumor activity of hydroxychloroquine with hormonal therapy with clinical benefit rate (CBR). Clinical benefits are defined as complete remission (CR), partial remission (PR) and stable disease (SD) | 18 months
  The anti-tumor activity of hydroxychloroquine with hormonal therapy with clinical benefit rate (CBR). Clinical benefits are defined as complete remission (CR), partial remission (PR) and stable disease (SD)
The disease-free survival (DFS) when adding hydroxychloroquine to hormonal therapy | 18 months
  The disease-free survival (DFS) when adding hydroxychloroquine to hormonal therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jiaxin Niu, MD, PhD, Principal Investigator — Western Regional Medical Center, Inc.
Locations (1):
- Western Regional Medical Center, Inc., Goodyear, Arizona, United States